CLINICAL TRIAL: NCT01399814
Title: Restricted Intravenous Fluid Regime Effects on Immunological Indicators of Elderly Patients Operated for Abdominal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Yu Wen Kui, Nanjing PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009NLY031
Record Dates: First submitted 2011-07-18; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2009-05

CONDITIONS: Surgery; Perioperative Care; Immunization; Abdominal Neoplasms
MeSH Terms: conditions — Abdominal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard fluid regimen group (Active Comparator): perioperative fluid treatment
  Interventions: Behavioral: perioperative fluid treatment
- restricted fluid regimen group (Experimental): perioperative fluid treatment
  Interventions: Behavioral: perioperative fluid management

INTERVENTIONS:
Behavioral: perioperative fluid management — No preloading of epidural analgesia,7ml/kg lactated ringer's solution was administered in first hour,and 5ml/kg.h during the following hours,and 1000ml of glucose 5% was administered on the rest of the day during operation.1000~1500ml crystalloid was administered on the days following operation
  Arms: restricted fluid regimen group
Behavioral: perioperative fluid treatment — 500 mL HAES 6% was accepted as preloading of epidural analgesia,12ml/kg.h lactated ringer's solution was administered during the operation ,and 1000ml of glucose 5% was administered on the rest of the day during operation.2000~2500ml crystalloid was administered on the days following operation
  Arms: standard fluid regimen group

SUMMARY:
The purpose of this study is to find out whether perioperative fluid restriction influence on postoperative immunological function. And discuss the probable mechanism that fluid restriction regime effect on clinical data.

DETAILED DESCRIPTION:
Perioperative fluid administration is a common therapy in clinical practice, and recent regime has a history about 50 years. Recently, clinicians found that traditional regime had some disadvantages, for example, pulmonary edema, increased cardiac load, increased body weight. And thus, perioperative fluid restriction regimen has been suggested and proved could reduce cardiopulmonary complications and mortality rates after major elective gastrointestinal surgery.

Patients were divided into two groups randomly and underwent restricted fluid regimen or traditional fluid regimen. We determined the complications and immunological function in two groups, and analyzed the relationship between complications and immunological changes. Based on this we decide the probable mechanism that perioperative fluid restriction effects on complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients(age≧65y) who was admitted for gastrointestinal cancer surgery were considered eligible if they had no life-threatening systemic disease (ASA groups 1~3)

Exclusion Criteria:

* lactation
* mental disorders
* language problems
* smoking within two weeks
* diabetes mellitus
* renal insufficiency
* disseminated cancer
* secondary cancers
* inflammatory bowel disease, or diseases hindering epidural analgesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 179 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
clinical perioperative complications | 30 days after surgery

SECONDARY OUTCOMES:
death | 30 days after surgery
adverse effects | 30 days after surgery
  ischemia and impairment of renal function